CLINICAL TRIAL: NCT04983524
Title: Evaluation of the Effect of Propolis Versus Calcium Hydroxide, Intracanal Medicaments on Post-Operative Pain in Patients With Necrotic Pulp (A Randomized Clinical Trial)
Brief Title: Propolis Versus Calcium Hydroxide on Post-Operative Pain in Patients With Necrotic Pulp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Serene Mohamed Hisham Sirry, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SSirry
Record Dates: First submitted 2021-07-11; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Post-Operative Pain, Chronic; Necrotic Pulp
Keywords: calcium hydroxide; propolis; post-operative pain; necrotic pulp
MeSH Terms: conditions — Pain, Postoperative; Dental Pulp Necrosis | interventions — Propolis; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis (Experimental): intervention intracanal medicament
  Interventions: Dietary Supplement: propolis
- Calcium Hudroxide (Active Comparator): Gold standard intracanal medicament
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Dietary Supplement: propolis — resinous product of honeybees
  Arms: Propolis
Drug: Calcium Hydroxide — Gold standard control intracanal medicament
  Arms: Calcium Hudroxide

SUMMARY:
Propolis is a resinous product of honeybees. Propolis is said to be effective against resistant microorganisms inside the root canal compared to the gold standard medication known as calcium hydroxide. The clinical trial tests the effect of propolis versus calcium hydroxide on pain in patients with necrotic teeth.

DETAILED DESCRIPTION:
Propolis is an immunomodulatory, antioxidant, flavonoid-rich resinous product of honeybees. Propolis was reported as less cytotoxic and more effective against resistant microorganisms than calcium hydroxide as well as biocompatible to the periradicular tissues than existing intracanal medicaments. The aim of this single-blinded randomized clinical trial was to evaluate the effect of propolis versus calcium hydroxide, intracanal medicaments, on post-operative pain in patients with necrotic single canal teeth. Methods: Forty-six participants with an age range of 20-40 years old, diagnosed as having necrotic pulp in their single-rooted, single canal teeth were included in this study, with 23 participants in each group. Treatment was done in two visits and intracanal medicament was applied for one week in between. Participants were instructed to rate their pain score by a numerical rating scale after 24, 48, 72 hours and at 7 days.

ELIGIBILITY:
Inclusion Criteria:

* • Asymptomatic patients with age range 20 - 40 years

  * Necrotic, single canal maxillary and mandibular teeth with periapical infection presented as radiolucency or widening in the periodontal membrane space.
  * Medically - free of any systemic disease
  * Teeth with complete root formation

Exclusion Criteria:

* • Pregnant or lactating females

  * Teeth with vital pulps, internal or external resorption or anatomic abnormalities
  * Teeth with cracks, curvatures, root caries and calcified canals
  * Double or triple-rooted teeth
  * Patients with facial swelling, acute pulpal or periapical lesion
  * Teeth that are not indicated for endodontic treatment: Bad oral hygiene, mobile or recessed
  * Previously endodontically-treated teeth

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
post-operative pain | one week. line of 10 points
  Categorical data on numerical rating scale

IPD SHARING:
Plan to Share IPD: Yes
the study protocol can be shared.
Supporting Information: Study Protocol
Time Frame: Will be available by November 2021
Access Criteria: will be uploaded on google drive